CLINICAL TRIAL: NCT04145180
Title: 3C-CUIDATE: Efectividad de un Programa de Recuperación Física en el Tratamiento de Las Secuelas Musculoesqueléticas, Funcionales y de Calidad de Vida en Pacientes de Cáncer de Cabeza y Cuello.
Brief Title: Effectiveness of a Physical Recovery Program for Head and Neck Cancer Patients (3C-CUIDATE)
Acronym: 3C-CUIDATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Carolina Fernández Lao, Dr. Carolina Fernández-Lao, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0045-N-16
Record Dates: First submitted 2019-10-09; First posted 2019-10-30 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer; Pain; Dysfunction
Keywords: Pain; Function; Quality of Life; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Therapy (Experimental): Manual Therapy-based intervention
  Interventions: Other: Manual therapy
- Control (No Intervention): Patients waiting list

INTERVENTIONS:
Other: Manual therapy — 40 minutes of physiotherapy, based on manual therapy sessions over 6 weeks. Three times a week.
  Arms: Manual Therapy

SUMMARY:
People receiving a head and neck cancer treatment often do not find an adequate therapeutic response for the side effects derived from this treatment. The objective of this study is to assess the effectiveness of a physical recovery program based on manual therapy over these problems.

Previous studies have shown the effectiveness of this type of programs on patients who have had cancer in other locations with clinically relevant results. There is a shortage of proposals for this subgroup of patients that require special attention. This project intends to carry out an experimental randomized controlled study with 84 patients treated of head and neck cancer who will be assigned randomly to the study groups: a) manual therapy program or, b) control group. The assessment refers to a baseline form (at the beginning of the study), at 6 weeks and at 6 months of patient follow-up.

DETAILED DESCRIPTION:
Manual therapy program consists of 3 sessions a week during 6 weeks, with a total of 18 appointments. Measurements are done before starting, after the last intervention and 6 months after finishing the treatment.

ELIGIBILITY:
Inclusion Criteria:

* To have ended their treatment in the previous 6-24 months
* To have no metastasis or active cancer
* To have cervical and/or temporomandibular joint pain >3 in a Visual Analogue Scale

Exclusion Criteria:

* Mental or physical illness preventing subjects from participating in the study
* Previous chronic pain conditions
* Previous cervical or temporomandibular joint pain
* Previous dysphagia disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 6 weeks
  Questionnaire EORTC QLQ-C30 was used for measuring quality of life
Health-related quality of life - 2 | 6 weeks
  Questionnaire EORTC QLQ-H&N-35 was used for measuring quality of life specifically in survivors of head and neck cancer
Pain Intensity | 6 weeks
  Visual Analogue Scale was used for evaluating pain intensity at cervical, temporomandibular joint, face and shoulder levels bilaterally.
  This consisted of a 10 cm horizontal line with the words "no pain" at the left extreme (0) and "pain as bad as it could be" at the right extreme (10)
Pressure pain thresholds | 6 weeks
  Pressure algometry (Force Dial DFK 20 analogue algometer, Wagner, Greenwich, USA) was assessed over the temporalis, masseter, upper trapezius and levator scapulae muscles and the C5-C6 zygapophyseal joint, the sternoclavicular joint and the tibialis anterior muscle as a distant reference muscle.
Shoulder and cervical active range of motion | 6 weeks
  Shoulder active range of motion (AROM) was assessed with a two-arms goniometer joined by a 360º protractor with the patient lying on a supine position. Cervical AROM was measured in a upright sitting position with a range of motion instrument (Performance Attainment Associates, Spine Products)

SECONDARY OUTCOMES:
Shoulder pain and disability perception | 6 weeks
  Shoulder pain and disability index (SPADI) was used to evaluate pain and disability perception of the patients at shoulder level.
Isometric handgrip strength | 6 weeks
  A digital dynamometer with adjustable grip (TKK 5101 Grip-D; Takei, Tokyo, Japan) was used to assess handgrip strength. Patients were standing in a upright position with the elbow in complete extension. Test was performed 3 times per hand, alternating both hands, with a 1-minute rest between trials.
Deep cervical flexors endurance | 6 weeks
  Endurance of deep cervical flexor muscles was assessed with the deep cervical flexor endurance test, with the patient in a supine lying position with the examiner's hands under his/her head and being told to fold the chin completely to the sternum and raising the head as minimum as possible without touching examiner's hands. Time is counted from when the patient lift his/her head until when he/she can no longer maintain the position.
Physical Fitness | 6 weeks
  International Fitness Scale (IFIS) was used to evaluate perceived physical fitness. It contains 4 physical fitness elements (cardiorespiratory endurance, muscular strength, speed/agility and flexibility) to categorize into 5 options, from very poor to very good
Maximal mouth opening | 6 weeks
  Mouth opening was evaluated with a sliding calliper measuring the inter-incisor distance asking the patients to open the mouth as maximum as possible
Temporomandibular disorders | 6 weeks
  The presence of temporomandibular disorders (TMD) was assessed with the Fonseca Anamneses Index, that classifies TMD as no dysfunction, light dysfunction, moderate dysfunction or severe dysfunction
Perceived fatigue | 6 weeks
  Piper Fatigue Scale - revised (PFS-r) was used to measure fatigue perception in head and neck cancer patients. It consists of 22 items divided into 4 subscales: behaviour, affection, emotional and cognitive. Each item is evaluated in a Visual Analogue Scale ranging from 0 to 10.
Fatigue | 6 weeks
  Fatigue perceived at the assessment moment was measured with a Visual Analogue Scale ranging from 0)no fatigue to 10) maximum fatigue perceived
Sleep quality | 6 weeks
  To evaluate sleep quality, Pittsburgh Sleep Quality Index (PSQI) was the instrument used. It consists of 19 self-rated questions related to sleep quality, including estimates of sleep duration and latency and the frequency and severity of specific sleep-related problems.
Sleeping disorders | 6 weeks
  Sleeping disorders were evaluated with a Visual Analogue Scale rating from 0)no disturbances to 10)impossible to sleep
Anxiety | 6 weeks
  Perception of anxiety at the assessment moment was measured with a Visual Analogue Scale rating from 0)no anxiety to 10)maximum anxiety perceived
Swallowing function | 6 weeks
  Eating Assessment Tool (EAT-10) was used to evaluate self-reported swallowing impairments. It is a 5 point Likert scale rating from no impairment to severe problem. The sum of all items contained on the questionnaire is used as the overall score, suggesting an abnormal swallowing when score is higher than 3
Swallowing difficulty | 6 weeks
  A Visual Analogue Scale was used to register swallowing difficulties, ranging from 0)no problems to 10)impossible to swallow

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Fernández-Lao, PhD, Study Chair — Universidad de Granada
Locations (1):
- Carolina Fernández Lao, Granada, Spain

REFERENCES:
- [Background] De Groef A, Van Kampen M, Vervloesem N, Dieltjens E, Christiaens MR, Neven P, Vos L, De Vrieze T, Geraerts I, Devoogdt N. Effect of myofascial techniques for treatment of persistent arm pain after breast cancer treatment: randomized controlled trial. Clin Rehabil. 2018 Apr;32(4):451-461. doi: 10.1177/0269215517730863. Epub 2017 Sep 15. PMID 28914087
- [Background] Sheikh A, Shallwani H, Ghaffar S. Postoperative shoulder function after different types of neck dissection in head and neck cancer. Ear Nose Throat J. 2014 Apr-May;93(4-5):E21-6. PMID 24817237
- [Background] Oz B, Memis A. Development of musculoskeletal complaints and functional disabilities in patients with laryngeal carcinoma after neck dissection sparing spinal accessory nerve. Eur J Cancer Care (Engl). 2009 Mar;18(2):179-83. doi: 10.1111/j.1365-2354.2008.00950.x. No abstract available. PMID 19267734
- [Background] Binczak M, Navez M, Perrichon C, Blanchard D, Bollet M, Calmels P, Couturaud C, Dreyer C, Espitalier F, Testelin S, Albert S, Moriniere S; SFORL Work Group. Management of somatic pain induced by head-and-neck cancer treatment: definition and assessment. Guidelines of the French Oto-Rhino-Laryngology- Head and Neck Surgery Society (SFORL). Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Sep;131(4):243-7. doi: 10.1016/j.anorl.2014.07.003. Epub 2014 Aug 6. PMID 25108356
- [Background] Cantarero-Villanueva I, Fernandez-Lao C, Fernandez-de-Las-Penas C, Lopez-Barajas IB, Del-Moral-Avila R, de la-Llave-Rincon AI, Arroyo-Morales M. Effectiveness of water physical therapy on pain, pressure pain sensitivity, and myofascial trigger points in breast cancer survivors: a randomized, controlled clinical trial. Pain Med. 2012 Nov;13(11):1509-19. doi: 10.1111/j.1526-4637.2012.01481.x. Epub 2012 Sep 7. PMID 22958507
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] van Wilgen CP, Dijkstra PU, van der Laan BF, Plukker JT, Roodenburg JL. Shoulder and neck morbidity in quality of life after surgery for head and neck cancer. Head Neck. 2004 Oct;26(10):839-44. doi: 10.1002/hed.20052. PMID 15390203
- [Background] Cardoso LR, Rizzo CC, de Oliveira CZ, dos Santos CR, Carvalho AL. Myofascial pain syndrome after head and neck cancer treatment: Prevalence, risk factors, and influence on quality of life. Head Neck. 2015 Dec;37(12):1733-7. doi: 10.1002/hed.23825. Epub 2014 Sep 25. PMID 24986588
- [Background] Sist T, Miner M, Lema M. Characteristics of postradical neck pain syndrome: a report of 25 cases. J Pain Symptom Manage. 1999 Aug;18(2):95-102. doi: 10.1016/s0885-3924(99)00054-8. PMID 10484856
- [Background] Gane EM, Michaleff ZA, Cottrell MA, McPhail SM, Hatton AL, Panizza BJ, O'Leary SP. Prevalence, incidence, and risk factors for shoulder and neck dysfunction after neck dissection: A systematic review. Eur J Surg Oncol. 2017 Jul;43(7):1199-1218. doi: 10.1016/j.ejso.2016.10.026. Epub 2016 Nov 17. PMID 27956321
- [Background] Gane EM, McPhail SM, Hatton AL, Panizza BJ, O'Leary SP. The relationship between physical impairments, quality of life and disability of the neck and upper limb in patients following neck dissection. J Cancer Surviv. 2018 Oct;12(5):619-631. doi: 10.1007/s11764-018-0697-5. Epub 2018 May 16. PMID 29770954